CLINICAL TRIAL: NCT06149234
Title: Effect Of Using Different Strips On Reducing The Most Common Error In Panoramic Imaging; Palatoglossal Air Space Shadow
Brief Title: Influencing Panoramic Imaging Errors With Strips
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasra Rahimipour (Other)
Responsible Party: Sponsor-Investigator, Kasra Rahimipour, Dr. Kasra Rahimipour, Tabriz University of Medical Sciences
Organization: Tabriz University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: TBZMED
Record Dates: First submitted 2023-11-14; First posted 2023-11-28 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Panoramic Radiography
Keywords: Panoramic Radiography,; Radiographic Error; Patient Positioning; Diagnostic Error; Palatoglossal Airspace Error

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: An oral and maxillofacial radiologist assessed the radiographs in single-blinded random selection to identify and record the errors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group (No Intervention): Normal panoramic positioning
- Fruit leather on the tongue (Experimental): The patient holding a stripe of fruit leather on the tongue while acquiring a panoramic image
  Interventions: Behavioral: Fruit leather on the tongue
- Chewing gum strip (Experimental): The patient holding a stripe of chewing gum on the tongue while acquiring a panoramic image
  Interventions: Behavioral: Chewing gum strip
- Celluloid matrix group (Experimental): The patient holding a stripe of celluloid matrix group on the tongue while acquiring a panoramic image
  Interventions: Behavioral: Celluloid matrix group

INTERVENTIONS:
Behavioral: Fruit leather on the tongue — The patient holds a fruit leather strip on the tongue while being exposed.
  Arms: Fruit leather on the tongue
Behavioral: Chewing gum strip — The patient holds a banana-tasting gum strip on the tongue while being exposed.
  Arms: Chewing gum strip
Behavioral: Celluloid matrix group — The patient holds a celluloid matrix stirp gum strip on the tongue while being exposed.
  Arms: Celluloid matrix group

SUMMARY:
Introduction: Panoramic radiography quality can be impaired by some errors such as positioning errors. Palatoglossal air space shadow error is one of the most common positioning errors and it's due to the tongue not sticking to the roof of the palate. Techniques used to deal with this error might help prevent unnecessary radiation to patients and save them time and money. The study aimed to investigate to investigate the effects of using celluloid matrix and edible tapes (fruit leather and chewing gum) on reducing the palatoglossal air space shadow error in panoramic imaging Methods: In our study, 270 patients referred to the Department of Radiology were randomised into three groups: a control group, a celluloid matrix group, and an edible tapes group. Before panoramic imaging, all patients were instructed to adhere their tongues to the roof of their mouths, with the distinction that for the celluloid matrix and edible tapes groups, patients were asked to place celluloid tapes, fruit leathers, or chewing gums on their tongues before doing so. The routine imaging process was then performed, and the results were compared across groups to evaluate the incidence of palatoglossal air space shadow error.

Results: *** Conclusion: ***

DETAILED DESCRIPTION:
Introduction Panoramic radiography is an extra-oral imaging technique and is considered an effective, fast, and relatively inexpensive diagnostic tool to examine dentofacial structures.Various errors such as open lips, shifted or tilted head position, inappropriate exposure parameters, movement of the patients, etc., have been reported for panoramic imaging, which reduce the quality of the images. The low quality of the radiographic images can result in misinterpretation by dentists, eventually leading to incorrect treatment plans. In addition, panoramic imaging errors ultimately can cause the repetition of radiography. In addition to wasting time and money, radiography repeating causes excess radiation exposure and increases the risk of potential damage in patients and medical radiation operators, including meningioma, brain tumors, and cancers, especially thyroid and Leukemia. Considering that the number of exposures to diagnostic radiation is relatively high during the lifetime, even a small increase related to the risk of cancer is of significant public importance.

Thus, numerous studies have highlighted the necessity of minimising medical and dental diagnostic radiation exposure as much as possible. Patient positional errors have been identified as the most frequent panoramic imaging errors, with some studies suggesting this is the case for nearly 95 percent of reported errors. Positional error and patient movement are two common reasons to reject dental imaging including intra-oral, extra-oral, and Cone-Beam Computed Tomography (CBCT). Thus, it is suggested that all dental radiography staff receive regular training focused on correct positioning techniques and reduction of patient movement.

The typical patient positioning errors in panoramic radiography include failure to rest the tongue against the palate, head positioned forward, head positioned backward, head twisted towards the left or right, head tilted to the left or right, the chin too high, the chin too low, a slumped position and inadequate neck extension, not resting the chin on the chin support, failing to use the bite guide, lips opened, patient movement during imaging and not removing the metal objects or prostheses. Among all the positional errors mentioned above, the most common error is the failure to keep the tongue against the palate.

Due to the failure of holding the tongue against the palate, the palatoglossal airspace (PGA) appears in panoramic radiographs as a dark radiolucent band under the hard palate and on the apices of the anterior maxillary teeth. This artefact significantly reduces the quality of the panoramic radiograph as it may be difficult or impossible to interpret the desired periapical region for correct diagnosis and treatment planning (for example, making it difficult to interpret cystic lesions in the anterior area of the upper jaw). In addition, when PGA falls on the ramus of the mandible, it may be mistaken for a fracture.

PGA may be seen unilaterally and asymmetrically as a localised radiolucent area if the patient swallows during panoramic imaging and momentarily does not touch the roof of the mouth. If the patient places only the tongue tip behind the maxillary teeth, a larger airspace is formed between the tongue and the hard palate.

As previous studies suggest, the average incidence of the error of not holding the tongue against the palate is nearly 40 percent. However, some studies have estimated that the frequency of this error in panoramic radiography can even reach 80-90 percent. Also, the tongue not being in contact with the palate is considered the most common error in the mixed dentition period. Overall, the incidence of positional errors, particularly the distance between tongue and palate, is reportedly higher in the mixed dentition period than in the permanent dentition period.

The main cause of PGA error is the patient's lack of understanding of the tongue-palate position and the radiography technicians' inability to clearly explain this issue to the patient and the lack of effective explanation and communication between the technician and the patient. During panoramic imaging, patients often cannot hold their tongue in a still position without moving, fully attached to the palate, and the technician cannot check that the patient has followed the instructions and that the tongue is in the correct position. Therefore, the operator should allocate sufficient time and use appropriate techniques to position the patient.

Although several studies have emphasised the importance and necessity of minimising PGA error, there is little research on the practical methods to achieve this goal.

It seems necessary to minimise the mentioned error using simple and practical techniques. In this regard, the present study evaluates the effect of using celluloid matrix tapes and oral tapes as a simple, and cheap method for proper positioning of the tongue on reducing the palatoglossal airway shadow error in panoramic imaging.

Materials and methods This study was conducted at the Oral and Maxillofacial Radiology Department, Faculty of Dentistry, Tabriz University of Medical Sciences, Iran, between 2021-09-29 and 2022-02-20. The study protocol was approved by the ethics committee of the university (Institutional Review Board: IR.TBZMED.REC.1399.730) Since there weren't similar studies to refer to, a pilot study was done with 30 patients from the oral and maxillofacial radiology department to figure out a suitable sample size. The patients were randomly divided and assessed in two groups of 15, each testing different materials: celluloid matrix tape and strips of food material. The initial results were promising, with a 99% success rate in the celluloid matrix tape group and 90% in the strips of food material group. Considering a Type I error of 0.05 and study power of 80%, 76 samples for each study group were calculated. To be on the safe side, this number was raised by an additional 20%, meaning 90 samples per group were used in the study. So, in total, the study worked with 270 samples, split evenly into three groups.

A total of 270 panoramic radiographs were acquired using a dental X-ray System (DR imaging system, RAYSCAN α-P, South Korea) according to the instructions of the manufacturer at 50/60 Hertz, 60-90 kW, 4-17 mA, and acquisition time of 14 s in the Scanner 2.0.1 software. The images were displayed and examined on an LCD (Liquid-Crystal Display) monitor (Dell E2014HF) with dimensions of 14.1 × 6.5 × 18.7 inches and a pixel pitch of 0.27 millimeters.

In this experimental study, all panoramic images were taken by a technician according to the patient positioning standards. The exposure settings were selected based on the patient's size and weight.

The main inclusion criterion was age above 15 years. Patients with a history of trauma, lesion, swelling, disseminated infection, physical and mental disabilities, severe gag reflex, cleft palate, difficulty in speech and tongue movement, allergy to the materials used in this study, and those reluctant to cooperate were excluded from the study.

The patients were randomised into three groups. Ninety patients received celluloid matrix strips of transparent polyester (Maquira Dental Products, Maringá, Brazil) with a 10 mm width and 30 mm length. In the second group, ninety patients were given edible strips. They were divided into two subgroups of 45 people. 45 patients received 10 × 30 mm strips of either commercial chewing gum (Banana Orion) with sweet banana flavor and 45 patients received sour fruit leather. Finally, as the third group, 90 patients were selected as the control group without giving any specific instructions.

Instruction of patients:

Panoramic imaging was carried out in the control group without any intervention (except for as a routine procedure, all of the patients in the control group were instructed to stick their tongue to the palate) and in accordance with the standard protocols of the Department of Oral and Maxillofacial Radiology.

Before panoramic imaging, the patients in edible and celluloid strip groups were instructed to put the given strips on their tongues. The strips were positioned in the anterior-posterior dimension at the middle third of the tongue, and in the transverse dimension in such a way that the centerline of the strip was placed in the central groove of the tongue. When adjusting the final head position in the machine, they were asked to elevate the strip to the roof of the mouth and hold it against the palate during the imaging procedure.

Assessment of radiographs An oral and maxillofacial radiologist assessed the radiographs in single-blinded random selection to identify and record the errors. The radiographs were classified as diagnostically acceptable, unacceptable, and excellent based on the degree of the palatoglossal air space shadow error.

Data analysis The statistical analyses were carried out using SPSSTM version 26 (IBM Corp., New York, NY; formerly SPSS Inc., Chicago, IL). The qualitative data were represented as frequency (percentage), and normal quantitative data were expressed as mean ± standard deviation. The Chi-square test compared the qualitative variables, and one-way analysis of variance (ANOVA) was used for quantitative variables with normal distribution. The intervention outcomes were evaluated using the logistic regression model. The differences with P<0.05 were considered statistically significant for all tests.

ELIGIBILITY:
Inclusion Criteria:

All patients over 15 years old attending the oral and maxillofacial department and are already prescribed for panoramic imaging.

Exclusion Criteria: Patients with a history of trauma, lesion, Swelling, disseminated infection, physical and mental disabilities, severe gag reflex, cleft palate, difficulty in speech and tongue movement, allergy to the materials used in this study, and those reluctant to cooperate were excluded from the study.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2022-03-20 (Actual)

PRIMARY OUTCOMES:
Investigating the panoramic images | 3 months
  Effect Of Using Different Strips On Reducing Palatoglossal Air Space Shadow: An oral and maxillofacial radiologist assessed the radiographs in single-blinded random selection to identify and record the errors. The radiographs were classified as diagnostically acceptable, unacceptable, and excellent based on the degree of the palatoglossal air space shadow error

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oral and Maxillofacial Surgery, Faculty of Dentistry, Tabriz University of Medical Sciences, Tabriz, Iran

IPD SHARING:
Plan to Share IPD: No